CLINICAL TRIAL: NCT02113956
Title: Harnessing the Power of Text Messaging to Invigorate AMSM HIV Preventive Behavior
Acronym: G2G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Northwestern University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00007481; 1R01MH096660-01A1 (NIH)
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: HIV
Keywords: HIV Prevention; Adolescent Men who Have Sex with Men (AMSM); Text-Messaging; Information-Motivation-Behavioral Skills(IMB)Model

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guy2Guy (G2G) (Experimental): G2G is a 6-week HIV prevention program delivered daily via text messaging to 14-18 year old males who self-identify as gay, bisexual, and/or queer. In addition to program content, participants are paired with another participant (i.e., a Text Buddy) with whom they can text throughout the program to provide support; and an on-demand advice line, G2Genie, which shares information about condoms, sex, relationships, and the lesbian, gay, bisexual, transgender (LGBT) community.
  Interventions: Behavioral: Guy2Guy (G2G)
- Healthy Lifestyle Control (No Intervention): The attention-matched control arm message content consists of information publicly available online related to living a healthy lifestyle. Content discussed includes: STD information, nutrition and sleep hygiene, self-esteem and body image, bullying, and drugs and alcohol. The control arm is 6-weeks in length (Week 6 is a review booster) and is delivered via text messaging. Messages are didactic and not tailored to user sexual experience. Additionally, the Text Buddy and G2Genie intervention program components are not available.

INTERVENTIONS:
Behavioral: Guy2Guy (G2G) — G2G is a text messaging-based healthy sexuality and HIV prevention program specifically for 14-18 year old GBQ adolescent males. Content is guided by the Information-Motivation-Behavioral Skills (IMB) model and focuses on: HIV information, motivations to engage in HIV preventive behavior, communication skills, behavioral skills (e.g., using a condom; HIV testing); and healthy/unhealthy relationships. Behavioral skills content is reinforced using brief online videos. The intervention is 5 weeks long. A "booster" is delivered 6-weeks post-intervention end and reviews the topics covered in the intervention. G2G content is tailored based upon whether one is abstinent or sexually active.
  Arms: Guy2Guy (G2G)

SUMMARY:
The purpose of this study is to examine whether Guy2Guy (G2G), a text messaging-based healthy sexuality and human immunodeficiency virus (HIV) prevention program intervention for 14-18 year gay, bisexual and queer men, is associated with HIV preventive behavior (e.g., condom use) compared to an attention-matched control group.

DETAILED DESCRIPTION:
Adolescent men who have sex with men (AMSM) are disproportionately affected by HIV. They account for almost 70% of HIV diagnoses among all young people and are the only risk group with an increasing number of HIV/AIDS diagnoses. Despite this disproportionate burden, current HIV prevention programs focus primarily on adults and heterosexual youth. As such, there is an urgent need for evidence-based HIV prevention programs targeting AMSM. Because issues affecting sexual health decisions among AMSM are unique, intervention programs cannot be translated from heterosexually focused interventions. Instead, they need to be designed from the ground up to ensure appropriately tailored content that resonates with the target population. Evidence-based HIV prevention programs targeting AMSM are urgently needed.

The Guy2Guy (G2G) intervention is a text messaging-based HIV prevention program designed for the specific needs of adolescent males who self-identify as gay, bisexual, or queer (GBQ) and are between the ages of 14-18 years. The intervention will be tested in a randomized controlled trial against an attention-matched control group which receives text messages about healthy lifestyle (e.g., exercise, nutrition). A total of 300 GBQ adolescent males will be into the study using an online recruitment strategy. The study is being conducted by researchers at the Center for Innovative Public Health Research and Northwestern University.

The primary efficacy outcome measures are unprotected sex acts and abstinence at 3-months follow-up. The investigators hypothesize that those in the G2G intervention will be significantly more likely to be engage in HIV preventive behavior (e.g., use condoms when having vaginal/anal sex) at 3-months follow-up compared to the attention-matched control group. Secondary efficacy outcomes include unprotected sex acts and abstinence at 3-month follow-up by sexual experience groups (i.e., ever had sex versus never had sex at baseline), HIV testing rates, and unprotected sex acts and abstinence at intervention end (5 weeks post enrollment) for those in the intervention versus control groups; and for participants who were sexually experienced and inexperienced at baseline, separately.

If effective, G2G has promise to be quickly and cost-effectively implemented to scale to help to curb the spread of HIV infection among AMSM long into adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as gay, bisexual, or queer
* Male biological sex
* Male gender
* Between the ages of 14-18
* English speaking
* Exclusive owners of a cell phone with an unlimited text messaging plan, have used text messaging for at least 6 months, and intend to have the same number for the next 6 months
* Able to provide informed assent, including an acceptable score on the "capacity to consent assessment"

Exclusion Criteria:

* Female or Transgender
* Participated in earlier study development activities

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Ybarra, PhD, Principal Investigator — Center for Innovative Public Health Research; Brian S Mustanski, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Center for Innovative Public Health Research, San Clemente, California
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prescott TL, Phillips Ii G, DuBois LZ, Bull SS, Mustanski B, Ybarra ML. Reaching Adolescent Gay, Bisexual, and Queer Men Online: Development and Refinement of a National Recruitment Strategy. J Med Internet Res. 2016 Aug 4;18(8):e200. doi: 10.2196/jmir.5602. PMID 27492781
- [Background] Ybarra ML, Prescott TL, Phillips GL 2nd, Parsons JT, Bull SS, Mustanski B. Ethical Considerations in Recruiting Online and Implementing a Text Messaging-Based HIV Prevention Program With Gay, Bisexual, and Queer Adolescent Males. J Adolesc Health. 2016 Jul;59(1):44-9. doi: 10.1016/j.jadohealth.2016.03.020. Epub 2016 May 13. PMID 27185621
- [Background] Phillips G 2nd, Ybarra ML, Prescott TL, Parsons JT, Mustanski B. Low Rates of Human Immunodeficiency Virus Testing Among Adolescent Gay, Bisexual, and Queer Men. J Adolesc Health. 2015 Oct;57(4):407-12. doi: 10.1016/j.jadohealth.2015.06.014. Epub 2015 Aug 26. PMID 26318671
- [Background] Ybarra ML, Prescott TL, Philips GL 2nd, Bull SS, Parsons JT, Mustanski B. Iteratively Developing an mHealth HIV Prevention Program for Sexual Minority Adolescent Men. AIDS Behav. 2016 Jun;20(6):1157-72. doi: 10.1007/s10461-015-1146-3. PMID 26238038
- [Background] DuBois LZ, Macapagal KR, Rivera Z, Prescott TL, Ybarra ML, Mustanski B. To have sex or not to have sex? An online focus group study of sexual decision making among sexually experienced and inexperienced gay and bisexual adolescent men. Arch Sex Behav. 2015 Oct;44(7):2027-40. doi: 10.1007/s10508-015-0521-5. Epub 2015 Apr 30. PMID 25925896
- [Background] Ybarra ML, DuBois LZ, Parsons JT, Prescott TL, Mustanski B. Online focus groups as an HIV prevention program for gay, bisexual, and queer adolescent males. AIDS Educ Prev. 2014 Dec;26(6):554-64. doi: 10.1521/aeap.2014.26.6.554. PMID 25490735
- [Background] Mustanski B, DuBois LZ, Prescott TL, Ybarra ML. A mixed-methods study of condom use and decision making among adolescent gay and bisexual males. AIDS Behav. 2014 Oct;18(10):1955-69. doi: 10.1007/s10461-014-0810-3. PMID 24906532
- [Result] Ybarra ML, Liu W, Prescott TL, Phillips G 2nd, Mustanski B. The Effect of a Text Messaging Based HIV Prevention Program on Sexual Minority Male Youths: A National Evaluation of Information, Motivation and Behavioral Skills in a Randomized Controlled Trial of Guy2Guy. AIDS Behav. 2018 Oct;22(10):3335-3344. doi: 10.1007/s10461-018-2118-1. PMID 29696403
- [Result] Ybarra ML, Prescott TL, Phillips GL 2nd, Bull SS, Parsons JT, Mustanski B. Pilot RCT Results of an mHealth HIV Prevention Program for Sexual Minority Male Adolescents. Pediatrics. 2017 Jul;140(1):e20162999. doi: 10.1542/peds.2016-2999. PMID 28659456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited through national advertisements on Facebook. Multiple ad images and text were used. To ensure a demographically representative sample, targeted ads were also used to enroll individuals from particular subgroups who are typically more difficult to engage in research
Groups:
- Guy2Guy (G2G): Guy2Guy (G2G) is a 6-week HIV prevention program delivered daily via text messaging to 14-18 year old males who self-identify as gay, bisexual, and/or queer. In addition to program content, participants were paired with another participant (i.e., a Text Buddy) with whom they can text throughout the program to provide support; and an on-demand advice line, G2Genie, which shares information about condoms, sex, relationships, and the LGBT (lesbian, gay, bisexual, transgender) community.
  Content is guided by the Information-Motivation-Behavioral Skills (IMB) model and focuses on: HIV information, motivations to engage in HIV preventive behavior, communication skills, behavioral skills (e.g., using a condom; HIV testing); and healthy/unhealthy relationships. Behavioral skills content was reinforced using brief online videos. The intervention is 5 weeks long. A "booster" is delivered 6-weeks post-intervention end and reviews the topics. Content is tailored by sexual experience.
- Healthy Lifestyle Control: The attention-matched control arm message content consists of information publicly available online related to living a healthy lifestyle. Content discussed includes: STD (sexual transmitted diseases) information, nutrition and sleep hygiene, self-esteem and body image, bullying, and drugs and alcohol. The control arm is 6-weeks in length (Week 6 is a review booster) and is delivered via text messaging. Messages are didactic and not tailored to user sexual experience. Additionally, the Text Buddy and G2Genie intervention program components are not available.
Period: Intervention End (5 Weeks Post Baseline)
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Started | 150 | 152
Completed | 141 | 148
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 4 | 3
Period: 3 Month Post-intervention
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Started | 141 | 148
Completed | 137 | 146
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Guy2Guy (G2G): Guy2Guy (G2G) is a 6-week HIV prevention program delivered daily via text messaging to 14-18 year old males who self-identify as gay, bisexual, and/or queer. In addition to program content, participants were paired with another participant (i.e., a Text Buddy) with whom they can text throughout the program to provide support; and an on-demand advice line, G2Genie, which shares information about condoms, sex, relationships, and the LGBT community.
  Content is guided by the Information-Motivation-Behavioral Skills (IMB) model and focuses on: HIV information, motivations to engage in HIV preventive behavior, communication skills, behavioral skills (e.g., using a condom; HIV testing); and healthy/unhealthy relationships. Behavioral skills content was reinforced using brief online videos. The intervention is 5 weeks long. A "booster" is delivered 6-weeks post-intervention end and reviews the topics. Content is tailored based upon whether one is abstinent or sexually active.
- Total: Total of all reporting groups
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control | Total
Number analyzed (Participants) | 150 | 152 | 302
Age, Customized [Count of Participants; unit: Participants]
  Age (y): 14 | 23 | 21 | 44
  Age (y): 15 | 37 | 33 | 70
  Age (y): 16 | 33 | 30 | 63
  Age (y): 17 | 36 | 23 | 59
  Age (y): 18 | 21 | 45 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 150 | 152 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 36 | 67
  Not Hispanic or Latino | 119 | 116 | 235
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 104 | 100 | 204
  Race: African American | 24 | 19 | 43
  Race: All other races | 22 | 33 | 55
Region of Enrollment [Number; unit: participants]
  United States | 150 | 152 | 302
Gay Identity [Count of Participants; unit: Participants] — Youth reported their sexual identity
  Participants | 114 | 105 | 219
Rural Setting [Count of Participants; unit: Participants] | 35 | 35 | 70
U.S. Region [Count of Participants; unit: Participants]
  Northeast | 20 | 26 | 46
  South | 47 | 53 | 100
  Midwest | 39 | 34 | 73
  West | 44 | 39 | 83
Family Income [Count of Participants; unit: Participants]
  Low Income | 33 | 42 | 75
  Middle Income | 88 | 73 | 161
  High Income | 29 | 37 | 66
Ever HIV Test [Count of Participants; unit: Participants] | 12 | 14 | 26
Sexually Inexperienced [Count of Participants; unit: Participants] | 73 | 76 | 149
Number of condomless sex acts [Mean (Standard Deviation); unit: number of condomless sex acts] | 1.3 (7.0) | 2.7 (9.9) | 2.02 (8.6)
Self-appraised greater than average or greater chances of getting HIV [Count of Participants; unit: Participants] | 47 | 47 | 94
Social Support [Mean (Standard Deviation); unit: units on a scale] — Multidimensional Scale of Perceived Social Support Total range: 0-36 Subscales for family, friends, and 'special person' are combined by summing Higher score is more positive social support
  units on a scale | 27.8 (9.4) | 27.9 (9.2) | 27.9 (9.3)
Self-esteem [Mean (Standard Deviation); unit: units on a scale] — Rosenberg Self-Esteem Scale Range: 0-30 Higher scores reflect higher self-esteem
  units on a scale | 19.3 (4.9) | 19.8 (4.7) | 19.6 (4.8)
Internalized stigma [Mean (Standard Deviation); unit: units on a scale] — Internalized Stigma Scale Range: 0-24 Higher scores reflect higher internalized stigma
  units on a scale | 5.9 (5.0) | 5.8 (5.2) | 5.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Condomless Sex Acts at 3-months Post-intervention
Description: The relative difference of unprotected anal and/or vaginal sex acts in the intervention versus control group at 3-months post-intervention. The count was truncated at 10 or higher to correct for over-dispersion.
Time Frame: 3-months post-intervention
Measure: Mean (Standard Deviation); unit: number of unprotected sex acts
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 137 | 146
number of unprotected sex acts | 2.85 (12.25) | 2.73 (15.97)
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Poisson regression; Incident Rate Ratio (IRR) = 1.42, 95% CI 2-sided [0.79 to 2.57] — Adjusted for age and baseline number of condomless sex acts

2. Primary Outcome: Percent of Boys Reporting Abstinence at 3-months Post-intervention
Description: At 3 months post intervention participants were asked whether or not they had had vaginal and anal sex in the past 90 days. Those who said no to both were coded as abstinent. The relative difference of abstinence (neither engaging in anal nor vaginal sex) was examined in the intervention versus control group.
Time Frame: 3-months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 137 | 146
Participants | 80 | 94
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.36 to 1.12]; Adjusted for age and baseline rate of abstinence

3. Secondary Outcome: Number of Unprotected Sex Acts Among Sexually Experienced at 3-months Post-intervention
Description: The relative difference of unprotected anal and/or vaginal sex acts in the intervention versus control group at 3-months post-intervention among youth who have ever had sex at baseline
Time Frame: 3-months post-intervention
Population: Youth who had ever had sex at baseline
Measure: Mean (Standard Deviation); unit: unprotected sex acts
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 69 | 71
unprotected sex acts | 5.48 (16.90) | 5.28 (22.66)
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Poisson; Incident Rate Ratio = .95, 95% CI 2-sided [0.45 to 2.02]; Adjusted for age and baseline number of condomless sex acts

4. Secondary Outcome: Number of Unprotected Sex Acts Among Sexually Inexperienced at 3-months Post-intervention
Description: The relative difference of unprotected anal and/or vaginal sex acts in the intervention versus control group at 3-months post-intervention among youth who have never had sex at baseline
Time Frame: 3-months post-intervention
Population: Youth who had never had sex at baseline
Measure: Mean (Standard Deviation); unit: unprotected sex acts
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 68 | 75
unprotected sex acts | .19 (.70) | .31 (1.43)
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Poisson; Incident Rate Ratio (IRR) = 0.62, 95% CI 2-sided [0.12 to 3.18]; Adjusted for age and baseline number of condomless sex acts

5. Secondary Outcome: Percent of Boys Reporting Abstinence Among Sexually Experienced at 3-months Post-intervention
Description: At 3 months post intervention participants were asked whether or not they had had vaginal and anal sex in the past 90 days. Those who said no to both were coded as abstinent. The relative difference of abstinence (neither engaging in anal nor vaginal sex) was examined among youth who have ever had sex at baseline in the intervention versus control groups.
Time Frame: 3-months post-intervention
Population: Youth who had ever had sex at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 69 | 71
Participants | 23 | 33
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.23 to 0.997]; Adjusted for age and baseline rate of abstinence

6. Secondary Outcome: Percent of Boys Reporting Abstinence Among Sexually Inexperienced at 3-months Post-intervention
Description: At 3 months post intervention participants were asked whether or not they had had vaginal and anal sex in the past 90 days. Those who said no to both were coded as abstinent. The relative difference of abstinence (neither engaging in anal nor vaginal sex) was examined among youth who have never had sex at baseline in the intervention versus control groups.
Time Frame: 3-months post-intervention
Population: Youth who had never had sex at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 68 | 75
Participants | 57 | 61
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.38 to 2.53]; Adjusted for age and baseline rate of abstinence

7. Secondary Outcome: Percent of Sexually Active Boys Reporting an HIV Test in the Past 3 Months at 3-months Post-intervention
Description: The relative difference of HIV testing over the past 3 months in the intervention versus control group at 3-months post-intervention among those who had ever vaginal or anal sex with a penis at baseline
Time Frame: 3-months post-intervention
Population: Youth who have ever had vaginal or anal sex with a penis at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 69 | 71
Participants | 38 | 20
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 3.42, 95% CI 2-sided [1.65 to 7.09]; Adjusted for age and baseline rate of HIV testing

8. Secondary Outcome: Number of Condomless Sex Acts at 5 Weeks Post-enrollment
Description: Relative difference of unprotected sex acts at intervention end (5 weeks post enrollment) for those in the intervention versus control groups
Time Frame: Intervention end (5-weeks post enrollment)
Measure: Mean (Standard Deviation); unit: unprotected sex acts
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 141 | 148
unprotected sex acts | 1.81 (8.94) | .89 (4.66)
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Poisson; Incident Risk Ratio (IRR) = 0.58, 95% CI 2-sided [0.22 to 1.5]; Adjusted for age and baseline number of condomless sex acts

9. Secondary Outcome: Percent of Boys Reporting Abstinence at 5 Weeks Post-enrollment
Description: The relative difference of abstinence (neither engaging in anal nor vaginal sex) in the intervention versus control group at intervention end (5 weeks post enrollment).
Time Frame: Intervention-end (5 weeks post-randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 141 | 148
Participants | 104 | 105
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.6 to 2.09]; Adjusted for age and baseline rate of abstinence

10. Secondary Outcome: Number of Unprotected Sex Acts Among Sexually Experienced Boys at 5 Weeks Post-enrollment
Description: The relative difference of unprotected anal and/or vaginal sex acts in the intervention versus control group intervention end (5 weeks post enrollment) among youth who have ever had sex at baseline
Time Frame: Intervention end (5-weeks post enrollment)
Population: Among the 144 youth who had ever had sex at baseline and completed the 5 week intervention end survey.
Measure: Mean (Standard Deviation); unit: unprotected sex acts
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 72 | 72
unprotected sex acts | 3.49 (12.31) | 1.76 (6.57)
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Incident Rate Ratio (IRR) = 0.6, 95% CI 2-sided [0.22 to 1.68]; Adjusted for age and baseline number of condomless sex acts

11. Secondary Outcome: Number of Unprotected Sex Acts Among Sexually Inexperienced Boys at 5 Weeks Post-enrollment
Description: The relative difference of unprotected anal and/or vaginal sex acts in the intervention versus control group at at intervention end (5 weeks post enrollment) among youth who have never had sex at baseline
Time Frame: Intervention end (5-weeks post enrollment)
Population: Among the 145 youth who had never had sex at baseline and completed the 5 week intervention end survey.
Measure: Mean (Standard Deviation); unit: unprotected sex acts
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 69 | 76
unprotected sex acts | 0.6 (.48) | .05 (.46)
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Incident Rate Ratio (IRR) = 1.10, 95% CI 2-sided [0.01 to 92.03]; Adjusted for age and baseline number of condomless sex acts

12. Secondary Outcome: Percent of Boys Reporting Abstinence Among Sexually Experienced at 5 Weeks Post-enrollment
Description: At 5 weeks post-enrollment, participants were asked whether or not they had had vaginal and anal sex since the beginning of the program. Those who said no to both were coded as abstinent. The relative difference of abstinence (neither engaging in anal nor vaginal sex) was examined among youth who have ever had sex at baseline in the intervention versus control groups.
Time Frame: Intervention end (5-weeks post enrollment)
Population: Among the 144 youth who had ever had sex at baseline and completed the 5 week intervention end survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 72 | 72
Participants | 37 | 36
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.46 to 1.88]; Adjusted for age and baseline rate of abstinence

13. Secondary Outcome: Percent of Boys Reporting Abstinence Among Sexually Inexperienced at 5 Weeks Post-enrollment
Description: At 5 weeks post-enrollment, participants were asked whether or not they had had vaginal and anal sex since the beginning of the program. Those who said no to both were coded as abstinent. The relative difference of abstinence (neither engaging in anal nor vaginal sex) was examined among youth who have never had sex at baseline in the intervention versus control groups.
Time Frame: Intervention end (5 weeks post enrollment)
Population: Among the 145 youth who had never had sex at baseline and completed the 5 week intervention end survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 69 | 76
Participants | 67 | 69
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 3.4, 95% CI 2-sided [0.88 to 16.95]; Adjusted for age and baseline rate of abstinence

14. Secondary Outcome: Percent of Sexually Experienced Boys Reporting Being Tested for HIV Since Program Start at 5 Weeks Post-enrollment
Description: The relative difference of HIV testing since the beginning of the program in the intervention versus control group at intervention end (5 weeks post enrollment) among those who ever had vaginal or anal sex with a penis at baseline
Time Frame: Intervention end (5 weeks post enrollment)
Population: Among the 144 youth who had ever had sex at baseline and completed the 5 week intervention end survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
Number analyzed (Participants) | 72 | 72
Participants | 28 | 13
Statistical Analysis 1: Comparison: Guy2Guy (G2G) vs Healthy Lifestyle Control; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.52 to 7.58]; Adjusted for age and baseline rate of HIV testing

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the study period (i.e., from baseline to 3-month follow-up)
Arm/Group | Guy2Guy (G2G) | Healthy Lifestyle Control
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/152
Other Adverse Events (participants affected / at risk) | 0/150 | 0/152

LIMITATIONS AND CAVEATS:
All data were collected via self-report questionnaires, so may be affected by recall and social desirability bias. The sample may not be representative of gay and bisexual youth who use the Internet less frequently or are not 'out' on social media.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2014-06-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02113956/ICF_000.pdf